CLINICAL TRIAL: NCT04107142
Title: A Phase I Dose-escalation Trial to Evaluate Haploidentical / Allogeneic Natural Killer Group 2D Ligand (NKG2DL)-Targeting Chimeric Antigen Receptor-grafted Gamma Delta (γδ) T Cells (CTM-N2D) in Subjects With Relapsed or Refractory Solid Tumour
Brief Title: Haplo / Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells for Relapsed or Refractory Solid Tumour
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CytoMed Therapeutics Pte Ltd (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CTM-N2D
Record Dates: First submitted 2019-09-21; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer; Triple Negative Breast Cancer; Sarcoma; Nasopharyngeal Carcinoma; Prostate Cancer; Gastric Cancer
Keywords: NKG2D; gamma; delta; T cell; CAR; chimeric antigen receptor; solid tumour; cancer immunotherapy; adoptive cell transfer
MeSH Terms: conditions — Colorectal Neoplasms; Triple Negative Breast Neoplasms; Sarcoma; Nasopharyngeal Carcinoma; Prostatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consisT of "3 + 3" dose escalation study design with 3 distinct dose level.
  The first dose level will be at 3 x 10^8 chimeric antigen receptor (CAR) grafted γδ T cells per infusion.
  The second dose level will be at 1 x 10^9 CAR-γδT cells per infusion. The third dose level will be increased to 3 x 10^9 cells CAR-γδT cells.
  Each cycle of therapy will consist of 4 intravenous infusions, given 7 days apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cell Therapy Group (Experimental): One arm study consisting of "3 + 3" dose escalation study design ranging from 3 x 10^8 - 3 x 10^9 cells CAR-γδ T cell.
  Each cycle of therapy will consist of 4 intravenous infusions, given 7 days apart.
  Interventions: Biological: Adoptive Cell Transfer of NKG2DL-targetting Chimeric Antigen Receptor-grafted Gamma Delta T cell

INTERVENTIONS:
Biological: Adoptive Cell Transfer of NKG2DL-targetting Chimeric Antigen Receptor-grafted Gamma Delta T cell — Adoptive Cell Transfer of Haploidentical / Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells (CTM-N2D)

SUMMARY:
This clinical trial is an open-label, single-centre, dose escalation, phase I study designed to investigate the safety and tolerability of Haploidentical / Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted Gamma Delta (γδ) T Cells (CTM-N2D) in Subjects with Relapsed or Refractory Solid Tumour. The study objectives of this phase I study are to determine the safety, activity and the safe dose of haploidentical or allogeneic NKG2DL-targeting chimeric antigen receptor-grafted γδ T cells given four times weekly in patients with relapsed or refractory solid tumors of different types.

DETAILED DESCRIPTION:
CTM-N2D-101 is a phase I dose-escalation study to evaluate the safety of CTM-N2D and the feasibility to produce CTM-N2D for three target dose levels between 3x10^8 - 3x10^9 per infusion will be tested. Four doses will be given at an interval of a week into subjects with relapsed or refractory solid tumors.

A typical 3+3 design will be used to determine the safe regimen basing on the incidence of dose-limiting toxicity (DLT). The identified safe regimen will be used for further phase II studies for selected indications.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old.
* Patient with specific cancer indications (see below).
* Disease must be measurable according to the corresponding guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or 2.
* Patient with adequate bone marrow reserve (Haemoglobin ≥10g/dl, Absolute Neutrophil Count (ANC)≥1,500/mm3, Platelet≥100,000/mm3), hepatic function (Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 3x upper limit of normal), renal function (serum creatinine < 120 µmol/L) and cardiac function (Left ventricular ejection fraction of ≥50% by ECHO).
* Patient must already have a previous tumour biopsy to confirm the disease.
* Patient must agree to sign the informed consent form (ICF).

Cancer-specific inclusion criteria of subject:

* Colorectal cancer: A documented metastatic colorectal adenocarcinoma and having received, being intolerant to or being unfit for at least two prior standard cancer therapy regimens as part of their primary treatment regimen or part of their treatment for management of recurrent/persistent disease.
* Breast cancer: A metastatic triple-negative breast cancer and having received at least two prior cancer therapy regimens as part of their treatment for management of recurrent/persistent disease.
* Sarcoma, nasopharyngeal cancer, prostate cancer or gastric cancer: A metastatic cancer and having received at least two prior cancer therapy regimens as part of their treatment for management of recurrent/persistent disease.

Exclusion Criteria:

* Patients with a tumour metastasis in the central nervous system.
* Patients who receive or are to receive any investigational product within the 4 weeks before the planned day for the first CTM-N2D administration.
* Patients who receive or are to receive chemotherapy within the 8 weeks before the planned day for the first CTM-N2D administration.
* Patients who are planned to receive concurrent growth factor, systemic steroid or other immunosuppressive therapy or cytotoxic agent.
* Patients who underwent major surgery within 4 weeks before the planned day for the first CTM-N2D administration.
* Patients who have active infections necessitating the use of antibiotics/antivirals treatment.
* Patients with a history of autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 6 months
  The primary endpoint of this dose-escalation study will be the occurrence of dose-limiting toxicities (DLTs) during 4 cycles of treatment and the week after treatment.

SECONDARY OUTCOMES:
Occurence of adverse events during therapy | 6 months
  A secondary outcome is to observe for the occurence of any adverse events (AEs) and serious adverse events (SAEs) during 4 cycles of treatment and the week after treatment
Observation of clinical efficacy | 6 months to 2 years
  A secondary outcome is to observe for the occurrence of objective clinical response at d31, M3, M6, M9, M12, M18 and M24 after the start of 1st cycle of treatment (assessed according to RECIST criteria, version 1.1)
Observation for progression-free survival | up to 2 years
  A secondary outcome is to observe for progression-free survival (PFS) and after the start of 1st cycle of treatment
Observation for duration of response | Up to 2 years
  A secondary outcome is to observe the duration of response in patients with objective response up to M24, After the start of 1st cycle of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Landmark Medical Centre, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No